CLINICAL TRIAL: NCT06077344
Title: WALANT in Ankle Fractures (Wide-Awake Local) Anesthesia No Tourniquet) and Applied Under Spinal Anesthesia Comparison of Clinical Results of Surgical Treatment; Randomized Prospective Clinical Research
Brief Title: WALANT and Spinal Anesthesia Comparison of Clinical Result in Ankle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, oguzhan albayrak, Medical Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: E-29624016-050.99-1682710
Record Dates: First submitted 2023-04-15; First posted 2023-10-11 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wide - Awake Local Anesthesia No Tourniquet (Active Comparator): WALANT solution used in our institution is prepared by mixing 20 ml of 2% lidocaine, with 0,4 ml 1:1000 (1 mg/ml) adrenaline in addition to 20 ml of 0,9% normal saline as described by Barros
  In the study, perop parameters to be checked are perop Visual Analogue Scale (VAS; at regular intervals (every 15 minutes, etc.) VAS evaluation, the highest value will be recorded), the time spent in the operating room
  Early postoperative parameters; Morphine consumption in PCA (in PCA device) the amount of morphine used in the postoperative 24 hours), the postoperative VAS (the postoperative 24th hour VAS) evaluation;).
  Interventions: Procedure: WALANT in Ankle Fractures (Wide-Awake Local) Anesthesia No Tourniquet) and Applied Under Spinal Anesthesia Comparison of Clinical Results of Surgical Treatment;ANT Procedure comparation
- Applied Under Spinal Anesthesia (Active Comparator): Applied Under Spinal Anesthesia
  Early postoperative parameters; Morphine consumption in PCA (in PCA device) the amount of morphine used in the postoperative 24 hours), the postoperative VAS (the postoperative 24th hour VAS) evaluation;).
  Interventions: Procedure: Applied Under Spinal Anesthesia of Clinical Results of Surgical Treatment

INTERVENTIONS:
Procedure: WALANT in Ankle Fractures (Wide-Awake Local) Anesthesia No Tourniquet) and Applied Under Spinal Anesthesia Comparison of Clinical Results of Surgical Treatment;ANT Procedure comparation — WALANT in Ankle Fractures (Wide-Awake Local) Anesthesia No Tourniquet) and Applied Under Spinal Anesthesia Comparison of Clinical Results of Surgical Treatment;ANT Procedure comparation
  Other Names: jetokain/ Adrenalin 1 mg/1 ml Biosel Ampul/DROGSAN SODYUM BIKARBONAT 84 MG/ML IV.
  Arms: Wide - Awake Local Anesthesia No Tourniquet
Procedure: Applied Under Spinal Anesthesia of Clinical Results of Surgical Treatment — Applied Under Spinal Anesthesia of Clinical Results of Surgical Treatment
  Arms: Applied Under Spinal Anesthesia

SUMMARY:
The application of the WALANT technique for foot and ankle surgery (joint fusion, implant removal and tendon repair, etc.) is limited. In our study, using the WALANT technique for ARIF in ankle fractures. The effect of this application on clinical outcomes will be prospectively evaluated.

DETAILED DESCRIPTION:
In this prospective randomized controlled study, a 1-year follow-up of ankle fracture patients who underwent regional anesthesia and those who underwent WALANT will be performed. Planning is being made with a total of 50 patients from 25 patients each in the experimental and control groups. Patients over 18 years of age with isolated bimalleolar or trimalleolar (no fixation required for posterior malleolus fracture) ankle fracture will be included in the study at Istanbul University Istanbul Faculty of Medicine, Department of Orthopaedics and Traumatology. Parameters to be evaluated preop in the study; patient's age, gender, smoking, comorbidities if any, fracture mechanism (traffic accident, fall from height, sprain etc.), open/closed fracture (open fractures above grade 1 will not be included), fracture type (including isolated bimalleolar or trimalleolar fractures and AO classification of those involving medial and lateral malleolus), date of hospitalization, date of surgery, American Society of Anesthesiologists (ASA) and Amsterdam Preoperative Anxiety and Information Score (APAIS) scale, and type of anesthesia administered to the patient. The highest value will be recorded), time in the operating room (the time between the patient's entry into the operating room and the time between the completion of all procedures and exit from the operating room), operation time (the time between the start of the incision and the end of suturing), implant applied to the lateral malleolus (plate and screw +/- syndesmosis screw), implant applied to the medial malleolus (cannulated screw/ plate and screw/ zuggurtung), amount of bleeding (difference between the amount of fluid flushed and the amount of aspirate in the aspiration collection cup). The parameters to be looked at early postop are morphine consumption in PCA (the amount of morphine used in the PCA device in the postop 24 hours), postop VAS (postop 24th hour VAS assessment; it can also be looked at after PCA is removed), hospitalization (the time between hospitalization and discharge), cost (to be calculated on the invoices sent to the insurance company for each patient from hospital accounting; it can be done for the entire cost or only anesthesia costs can be compared). The parameters to be examined late postop will be; AOFAS (at 6 and 12 months), union status (the date when callus formation is seen in 3 of 4 cortices in AP and lateral radiographs in the patient's periodic controls will be accepted as the date of union), ipsilateral quadriceps diameter (measurement made from 1 or more than 1 thigh level at 6 and 12 months), contralateral quadriceps diameter (measurement made from 1 or more than 1 thigh level at 6 and 12 months).

ELIGIBILITY:
Inclusion Criteria:

->18 years

* Isolated bimalleolar ankle fracture
* Isolated trimalleolar ankle fracture (posterior malleolar fracture will not be operative)

Exclusion Criteria:

* < 18 years
* vasculitis
* Raynaud's disease
* Peripheral vascular disease
* peripheral neuropathy
* Lidocaine and epinephrine hypersensitivity
* Grade >1 open fractures
* Maisonneuve, talus and posterior malleolus (requires fixation) fractures
* multitrauma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Perop VAS | Perop
  VAS assessment at certain intervals (every 15 minutes, etc.), the highest value will be recorded
Postop Morphine Consume | 24 hours
  The amount of morphine used in the PCA device within 24 hours postop

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department Orthopaedics and Traumatology, Istanbul, Çapa / Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Fish MJ, Bamberger HB. Wide-Awake Local Anesthesia No Tourniquet (WALANT) Hand Surgery. 2023 Apr 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK570646/ PMID 34033408
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK570646/